CLINICAL TRIAL: NCT05581160
Title: Assess the Performance of Metagenomic Sequencing in the Diagnosis of STI (NGS-IST)
Acronym: NGS-IST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IMEA62
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2023-05

CONDITIONS: Sexually Transmitted Infections (Not HIV or Hepatitis); Chlamydia Trachomatis Infection; Neisseria Gonorrhoeae Infection; Mycoplasma Genitalium Infection
Keywords: Metagenomics Next-Generation-Sequencing (NGS); Sexually Transmitted Infections (STI); Pre-Exposure Prophylaxis (PrEP); Men who have Sex with Men (MSM)
MeSH Terms: conditions — Sexually Transmitted Diseases; Hepatitis; Gonorrhea; Homosexuality

STUDY DESIGN:
Intervention Model Description: 12-months prospective multicenter longitudinal cohort with the biological samples collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 12-months prospective multicenter longitudinal cohort with the biological samples collection. (Experimental): This is a single-arm interventional study. After acceptance of the study (signature of the informed consent form), patients are included in the single-arm interventional study for a period of 12 months with follow-up visits every 3 months and intermediate visits in the case of the symptoms presence or sexual contacts with partners having STIs (corresponding to standard care for the PrEP users).
  Interventions: Diagnostic Test: Assess the Performance of Metagenomic Sequencing in the Diagnosis of STI (NGS-IST)

INTERVENTIONS:
Diagnostic Test: Assess the Performance of Metagenomic Sequencing in the Diagnosis of STI (NGS-IST) — Proposal of the study to all eligible adult patients coming for pre-exposure prophylaxis (PrEP) consultations from the Infectious Diseases Department of Saint-Antoine and Tenon Hospitals (with delivery of a patient's information and signing an informed consent form).
  During each visit (D0, M3, M6, M9, M12 and intermediate visits), patients will be asked to:
  * Respond to a questionnaire on their history of taking antibiotics, STIs, their foreign travels, their consumption of tobacco, drugs, alcohol and their sexual practices.
  * Perform the following additional samples at each visit, including the intermediate: rectal and throat swabs, urine sample and swab from the lesions in the case of ulceration presence due to STIs.
  The diagnosis of STIs (NG and MG) will be carried out using 2 techniques: the reference technique and the Next-Generation-Sequencing (NGS) technique.
  A serum sample will be collected during routine care. All samples will be stored after the analysis under -80° C.

SUMMARY:
The main objective of the study will be to assess the performance of the Next-Generation-Sequencing (NGS) diagnostics of Chlamydia trachomatis and Neisseria gonorrhoeae compared to reference techniques.

DETAILED DESCRIPTION:
Sexually Transmitted Infections (STIs) have become a major global public health problem and are among the most common infections. The increase antibiotic resistance, particularly in Neisseria gonorrhoeae and Mycoplasma genitalium, is of concern. Currently, the diagnosis of STIs is based on specific tests by pathogen, mainly by standard culture allowing an antibiotic susceptibility testing, gene amplification tests possibly allowing the search for resistance genes and serologies.

Next-Generation-Sequencing (NGS) is based on the detection and analysis of any DNA and RNA present in the studied sample with a high degree of sensitivity, this method enables the precise identification of non-human sequences regardless its bacterial, viral or parasitologic origin, to detect resistance genes and to characterize the strains.

The investigators propose to assess the performance of NGS for the diagnosis of STIs. A cohort of 332 PrEP users from Saint-Antoine and Tenon Hospitals will be followed for this purpose every 3 months during 1 year (including also the intermediate visits if needed in case of STIs symptoms).

The main objective of the study will be to assess the performance of the NGS diagnostics of Chlamydia trachomatis and Neisseria gonorrhoeae compared to reference techniques.

The secondary objectives will be (i) to evaluate the performance of the diagnosis by NGS of the other STIs compared to the reference techniques, (ii) to evaluate the interest and the sensitivity of a 3 sites pooled sample "urine, throat and rectum" and the swab sampling from the ulcer lesions in the case of the ulcerations presence for the diagnosis of STIs, (iii) to describe the natural history of colonization with Mycoplasma genitalium and the appearance of resistance or pressure of antibiotic selection and (iv) to evaluate the prevalence of agents not usually sought in screening for STI (HSV-1, HSV-2, Haemophilus ducreyi, Campylobacter sp, Shigella sp, Clostridioides difficile, Entamoeba histolytica).

Improved diagnosis of STIs and resistance will allow a better patient management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* MSM
* PrEP users
* Acceptance of study constraints
* With or without Social Security scheme or State Medical Aid
* Signature of consent form to participate in the study

Exclusion Criteria:

* Language barrier making questioning impossible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men who have sex with men (MSM).
Enrollment: 332 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
To evaluate the performance of NGS metagenomic diagnosis of Chlamydia trachomatis (Ct) and Neisseria gonorrhoeae (Ng) compared to reference techniques. | 12 months
  Sensitivity, specificity, positive and negative predictive values of NGS compared to reference techniques for Ng and Ct.

SECONDARY OUTCOMES:
To evaluate the performance of the diagnosis by NGS of the other STIs compared to the reference techniques. | 12 months
  Sensitivity, specificity, positive and negative predictive values of NGS compared to reference techniques for other sexually transmitted infections (STIs).
Describe the epidemiology of circulating strains by molecular typing. | 12 months
  Total number of cases of Ct, Ng, agents not usually screened for in STI screening compared to the number of subjects at the time of their inclusion in the study cohort, with 95% confidence interval.
Estimate the incidence and describe the natural history of colonization by Mycoplasma genitalium (Mg). | 12 months
  Number of new cases Mycoplasma genitalium (Mg) compared to the number of subjects followed in the study cohort per month of follow-up.
Estimate the incidence of the appearance of Mycoplasma genitalium resistance under antibiotic selection pressure. | 12 months
  Number of new cases Mycoplasma genitalium (Mg) compared to the number of subjects followed in the study cohort per month of follow-up under antibiotic selection pressure.
Characterize circulating Neisseria gonorrhoeae (Ng) clones. | 12 months
  Total number of cases of circulating Neisseria gonorrhoeae (Ng) clones compared to the number of subjects at the time of their inclusion in the study cohort, with 95% confidence interval.
Characterize the circulating serotypes of Chlamydia trachomatis (Ct). | 12 months
  Total number of cases of circulating serotypes of Chlamydia trachomatis (Ct) compared to the number of subjects at the time of their inclusion in the study cohort, with 95% confidence interval.
Estimate the incidence of agents not usually screened for in STI screening (HSV-1, HSV-2, HPV, Mycoplasma hominis, Ureaplasma sp, Haemophilus ducreyi, Campylobacter sp, Shigella sp, Clostridium difficile, Entamoeba histolytica). | 12 months
  Number of new cases of agents not usually tested for in STI screening compared to the number of subjects followed in the study cohort per month of follow-up.
Determine the factors associated with STI events. | 12 months
  Hazard ratio of determinants (factors) associations with the STI cases incidence.

CONTACTS AND LOCATIONS:
Overall Officials: Karine Lacombe, Pr, PhD, Study Chair — IPLESP INSERM UMR-S1136; Laure Surgers, MD, Principal Investigator — Service des Maladies Infectieuses et Tropicales Hôpital Saint-Antoine; Martin Siguier, MD, Principal Investigator — Service des Maladies Infectieuses et Tropicales et Tenon Hôpital; Christophe Rodriguez, MD, Study Director — INSERM U955 Eq18 CHU Henri Mondor
Locations (2):
- France (2):
  - Service des Maladies Infectieuses et Tropicales Hôpital Saint-Antoine, Paris
  - Service des Maladies Infectieuses et Tropicales Hôpital Tenon, Paris

IPD SHARING:
Plan to Share IPD: No
Will be decided later by the scientific committee at the end of the study.

REFERENCES:
- [Background] Abdool Karim Q, Abdool Karim SS, Frohlich JA, Grobler AC, Baxter C, Mansoor LE, Kharsany AB, Sibeko S, Mlisana KP, Omar Z, Gengiah TN, Maarschalk S, Arulappan N, Mlotshwa M, Morris L, Taylor D; CAPRISA 004 Trial Group. Effectiveness and safety of tenofovir gel, an antiretroviral microbicide, for the prevention of HIV infection in women. Science. 2010 Sep 3;329(5996):1168-74. doi: 10.1126/science.1193748. Epub 2010 Jul 19. PMID 20643915
- [Background] Chaix ML, Charreau I, Pintado C, Delaugerre C, Mahjoub N, Cotte L, Capitant C, Raffi F, Cua E, Pialoux G, Tremblay C, Meyer L, Molina JM; ANRS IPERGAY Study Group. Effect of On-Demand Oral Pre-exposure Prophylaxis With Tenofovir/Emtricitabine on Herpes Simplex Virus-1/2 Incidence Among Men Who Have Sex With Men: A Substudy of the ANRS IPERGAY Trial. Open Forum Infect Dis. 2018 Nov 8;5(11):ofy295. doi: 10.1093/ofid/ofy295. eCollection 2018 Nov. PMID 30539039
- [Background] Deschamps O, Ortonne N, Hue S, Rodriguez C, Deschodt C, Hirsch G, Colin A, Gregoire L, Delfau-Larue MH, Chosidow O, Wolkenstein P, Ingen-Housz-Oro S. Acute exanthemas: a prospective study of 98 adult patients with an emphasis on cytokinic and metagenomic investigation. Br J Dermatol. 2020 Feb;182(2):355-363. doi: 10.1111/bjd.18166. Epub 2019 Aug 9. PMID 31127953
- [Background] Fourati S, Rodriguez C, Hezode C, Soulier A, Ruiz I, Poiteau L, Chevaliez S, Pawlotsky JM. Frequent Antiviral Treatment Failures in Patients Infected With Hepatitis C Virus Genotype 4, Subtype 4r. Hepatology. 2019 Feb;69(2):513-523. doi: 10.1002/hep.30225. Epub 2019 Jan 5. PMID 30125371
- [Background] Hernando Rovirola C, Spiteri G, Sabido M, Montoliu A, Gonzalez V, Casabona J, Cole MJ, Noori T, Unemo M. Antimicrobial resistance in Neisseria gonorrhoeae isolates from foreign-born population in the European Gonococcal Antimicrobial Surveillance Programme. Sex Transm Infect. 2020 May;96(3):204-210. doi: 10.1136/sextrans-2018-053912. Epub 2020 Feb 4. PMID 32019895
- [Background] Hoornenborg E, Coyer L, Achterbergh RCA, Matser A, Schim van der Loeff MF, Boyd A, van Duijnhoven YTHP, Bruisten S, Oostvogel P, Davidovich U, Hogewoning A, Prins M, de Vries HJC; Amsterdam PrEP Project team in the HIV Transmission Elimination AMsterdam (H-TEAM) Initiative. Sexual behaviour and incidence of HIV and sexually transmitted infections among men who have sex with men using daily and event-driven pre-exposure prophylaxis in AMPrEP: 2 year results from a demonstration study. Lancet HIV. 2019 Jul;6(7):e447-e455. doi: 10.1016/S2352-3018(19)30136-5. Epub 2019 Jun 6. PMID 31178284
- [Background] Looker KJ, Elmes JAR, Gottlieb SL, Schiffer JT, Vickerman P, Turner KME, Boily MC. Effect of HSV-2 infection on subsequent HIV acquisition: an updated systematic review and meta-analysis. Lancet Infect Dis. 2017 Dec;17(12):1303-1316. doi: 10.1016/S1473-3099(17)30405-X. Epub 2017 Aug 23. PMID 28843576
- [Background] Molina JM, Charreau I, Chidiac C, Pialoux G, Cua E, Delaugerre C, Capitant C, Rojas-Castro D, Fonsart J, Bercot B, Bebear C, Cotte L, Robineau O, Raffi F, Charbonneau P, Aslan A, Chas J, Niedbalski L, Spire B, Sagaon-Teyssier L, Carette D, Mestre SL, Dore V, Meyer L; ANRS IPERGAY Study Group. Post-exposure prophylaxis with doxycycline to prevent sexually transmitted infections in men who have sex with men: an open-label randomised substudy of the ANRS IPERGAY trial. Lancet Infect Dis. 2018 Mar;18(3):308-317. doi: 10.1016/S1473-3099(17)30725-9. Epub 2017 Dec 8. PMID 29229440
- [Background] Nieuwenhuis RF, Ossewaarde JM, Gotz HM, Dees J, Thio HB, Thomeer MG, den Hollander JC, Neumann MH, van der Meijden WI. Resurgence of lymphogranuloma venereum in Western Europe: an outbreak of Chlamydia trachomatis serovar l2 proctitis in The Netherlands among men who have sex with men. Clin Infect Dis. 2004 Oct 1;39(7):996-1003. doi: 10.1086/423966. Epub 2004 Sep 8. PMID 15472852
- [Background] Ong JJ, Baggaley RC, Wi TE, Tucker JD, Fu H, Smith MK, Rafael S, Anglade V, Falconer J, Ofori-Asenso R, Terris-Prestholt F, Hodges-Mameletzis I, Mayaud P. Global Epidemiologic Characteristics of Sexually Transmitted Infections Among Individuals Using Preexposure Prophylaxis for the Prevention of HIV Infection: A Systematic Review and Meta-analysis. JAMA Netw Open. 2019 Dec 2;2(12):e1917134. doi: 10.1001/jamanetworkopen.2019.17134. PMID 31825501
- [Background] Rodriguez C, Jary A, Hua C, Woerther PL, Bosc R, Desroches M, Sitterle E, Gricourt G, De Prost N, Pawlotsky JM, Chosidow O, Sbidian E, Decousser JW; Multidisciplinary Necrotizing Fasciitis Study Group. Pathogen identification by shotgun metagenomics of patients with necrotizing soft-tissue infections. Br J Dermatol. 2020 Jul;183(1):105-113. doi: 10.1111/bjd.18611. Epub 2019 Dec 2. PMID 31610037
- [Background] Rodriguez C, Gricourt G, Ndebi M, Demontant V, Poiteau L, Burrel S, Boutolleau D, Woerther PL, Calvez V, Stroer S, Pawlotsky JM. Fatal Encephalitis Caused by Cristoli Virus, an Emerging Orthobunyavirus, France. Emerg Infect Dis. 2020 Jun;26(6):1287-1290. doi: 10.3201/eid2606.191431. PMID 32441621
- [Background] Sitterle E, Rodriguez C, Mounier R, Calderaro J, Foulet F, Develoux M, Pawlotsky JM, Botterel F. Contribution of Ultra Deep Sequencing in the Clinical Diagnosis of a New Fungal Pathogen Species: Basidiobolus meristosporus. Front Microbiol. 2017 Mar 7;8:334. doi: 10.3389/fmicb.2017.00334. eCollection 2017. PMID 28326064
- [Background] Unemo M, Shafer WM. Antimicrobial resistance in Neisseria gonorrhoeae in the 21st century: past, evolution, and future. Clin Microbiol Rev. 2014 Jul;27(3):587-613. doi: 10.1128/CMR.00010-14. PMID 24982323
- [Background] Van Praet JT, Steyaert S, Vandecasteele S, Van Den Bergh B, Mahieu H, De Buyser S, Grootaert V, Descheemaeker P, Reynders M. Mycoplasma genitalium acquisition and macrolide resistance after initiation of HIV pre-exposure prophylaxis in men who have sex with men. Sex Transm Infect. 2020 Sep;96(6):396-398. doi: 10.1136/sextrans-2019-054335. Epub 2020 Jan 2. PMID 31896737
- [Background] Wilson MR, Sample HA, Zorn KC, Arevalo S, Yu G, Neuhaus J, Federman S, Stryke D, Briggs B, Langelier C, Berger A, Douglas V, Josephson SA, Chow FC, Fulton BD, DeRisi JL, Gelfand JM, Naccache SN, Bender J, Dien Bard J, Murkey J, Carlson M, Vespa PM, Vijayan T, Allyn PR, Campeau S, Humphries RM, Klausner JD, Ganzon CD, Memar F, Ocampo NA, Zimmermann LL, Cohen SH, Polage CR, DeBiasi RL, Haller B, Dallas R, Maron G, Hayden R, Messacar K, Dominguez SR, Miller S, Chiu CY. Clinical Metagenomic Sequencing for Diagnosis of Meningitis and Encephalitis. N Engl J Med. 2019 Jun 13;380(24):2327-2340. doi: 10.1056/NEJMoa1803396. PMID 31189036
- [Background] Wilson MR, Naccache SN, Samayoa E, Biagtan M, Bashir H, Yu G, Salamat SM, Somasekar S, Federman S, Miller S, Sokolic R, Garabedian E, Candotti F, Buckley RH, Reed KD, Meyer TL, Seroogy CM, Galloway R, Henderson SL, Gern JE, DeRisi JL, Chiu CY. Actionable diagnosis of neuroleptospirosis by next-generation sequencing. N Engl J Med. 2014 Jun 19;370(25):2408-17. doi: 10.1056/NEJMoa1401268. Epub 2014 Jun 4. PMID 24896819
- [Background] Surgers L, Chiarabini T, Royer G, Rougier H, Mercier-Darty M, Decre D, Valin N, Woerther PL, Decousser JW, Girard PM, Lacombe K, Boyd A. Evidence of Sexual Transmission of Extended-Spectrum beta-Lactamase-Producing Enterobacterales: A Cross-sectional and Prospective Study. Clin Infect Dis. 2022 Oct 29;75(9):1556-1564. doi: 10.1093/cid/ciac218. PMID 35307740